CLINICAL TRIAL: NCT03030105
Title: A Randomized, Double-blind, Placebo-controlled, Single-dose, 6-Period Crossover Study to Evaluate the Effects of BPN14770 on Scopolamine-induced Cognitive Impairment in Healthy Volunteers
Brief Title: Study to Evaluate the Effects of BPN14770 on Scopolamine-induced Cognitive Impairment in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tetra Discovery Partners (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BPN14770-CNS-103
Record Dates: First submitted 2017-01-17; First posted 2017-01-24 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Alzheimer Disease
Keywords: Cognition; Dementia; Phosphodiesterase Type 4D; PDE4D; Scopolamine; Donepezil
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — BPN14770; Donepezil; Scopolamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- A) P:P:P (Placebo Comparator): Scopolamine placebo : BPN14770 placebo : Donepezil placebo
  Interventions: Drug: BPN14770 placebo; Drug: Donepezil placebo; Drug: Scopolamine placebo
- B) S:P:P (Placebo Comparator): Scopolamine 0.5mg : BPN14770 placebo : Donepezil placebo
  Interventions: Drug: BPN14770 placebo; Drug: Donepezil placebo; Drug: Scopolamine 0.6 MG/ML
- C) S:B:P (Experimental): Scopolamine 0.5mg : BPN14770 10mg : Donepezil placebo
  Interventions: Drug: BPN14770; Drug: Donepezil placebo; Drug: Scopolamine 0.6 MG/ML
- D) S:B:P (Experimental): Scopolamine 0.5mg : BPN14770 50mg : Donepezil placebo
  Interventions: Drug: BPN14770; Drug: Donepezil placebo; Drug: Scopolamine 0.6 MG/ML
- E) S:P:D (Active Comparator): Scopolamine 0.5mg : BPN14770 placebo : Donepezil 10mg
  Interventions: Drug: BPN14770 placebo; Drug: Donepezil; Drug: Scopolamine 0.6 MG/ML
- F) S:B:D (Experimental): Scopolamine 0.5mg : BPN14770 50mg : Donepezil 10mg
  Interventions: Drug: BPN14770; Drug: Donepezil; Drug: Scopolamine 0.6 MG/ML

INTERVENTIONS:
Drug: BPN14770 — investigational drug
  Arms: C) S:B:P; D) S:B:P; F) S:B:D
Drug: BPN14770 placebo — placebo
  Arms: A) P:P:P; B) S:P:P; E) S:P:D
Drug: Donepezil — comparator
  Other Names: Aricept
  Arms: E) S:P:D; F) S:B:D
Drug: Donepezil placebo — placebo
  Other Names: Aricept placebo
  Arms: A) P:P:P; B) S:P:P; C) S:B:P; D) S:B:P
Drug: Scopolamine 0.6 MG/ML — cognition impairment
  Other Names: Hyoscine s.c.
  Arms: B) S:P:P; C) S:B:P; D) S:B:P; E) S:P:D; F) S:B:D
Drug: Scopolamine placebo — placebo
  Other Names: Hyoscine s.c. placebo
  Arms: A) P:P:P

SUMMARY:
This is a Phase 1, randomized, double-blind, placebo-controlled, 6-period crossover study to evaluate the effects of BPN14770 10 mg and 50 mg in reversing scopolamine-induced cognitive impairment in healthy volunteers. A positive control, donepezil 10 mg, will be included, and additivity of BPN14770 50 mg to donepezil 10 mg in reversing scopolamine effects will also be evaluated.

DETAILED DESCRIPTION:
A total of 38 subjects will be enrolled into the study. The study duration will be up to 12 weeks with 6 weeks of single-dose Treatment Visits. The study will consist of a Screening Visit (up to 28 days prior to first study drug administration), six inpatient Treatment Visits (Periods 1 through 6), and a Follow-Up/Early Termination Visit (7-10 days after the last dose of study medication). An additional study visit may be necessary to complete the required cognitive test familiarization if not completed during the Screening Visit. Each Treatment Visit will occur approximately one week apart, allowing a 6 to 8 day washout period.

Subjects will be randomized to 1 of 6 treatment sequences based on a computer-generated randomization schedule. Subjects will receive all 6 treatments as specified by the treatment sequence according to a 6 × 6 Williams Latin square design. The following treatments will be administered:

A. Scopolamine placebo + BPN14770 placebo + donepezil placebo

B. Scopolamine 0.5 mg + BPN14770 placebo + donepezil placebo

C. Scopolamine 0.5 mg + BPN14770 10 mg + donepezil placebo

D. Scopolamine 0.5 mg + BPN14770 50 mg + donepezil placebo

E. Scopolamine 0.5 mg + donepezil 10 mg +BPN14770 placebo

F. Scopolamine 0.5 mg + BPN14770 50 mg + donepezil 10 mg

During each of the Treatment Visits (Periods 1 through 6), subjects will be admitted to the Clinical Research Unit (CRU) the day prior to each study drug administration (Day -1) and discharged the day after study drug administration (Day 2). On the morning of study drug administration (Day 1), subjects will be given study drug (BPN14770, donepezil, or placebo) with 240mL of room temperature water 2 hours prior to the scopolamine or scopolamine placebo sc injection. The timing for study drug administration will be referred to as t-2 (Hour -2). Breakfast should be available approximately 30 minutes following the morning drug administration. Two hours after study drug administration, the scopolamine or scopolamine placebo sc injection will be administered. The time at which the scopolamine or scopolamine placebo sc injection is administered will be referred to as t0 (Hour 0).

Cognitive testing will be performed 30 minutes prior to treatment with scopolamine injection and at hours 1, 2, 3, 4, and 6 post-scopolamine injection.

PK samples will be collected during the treatment period to confirm study drug is present.

Safety assessments throughout the study will include physical exams, ECGs, vital signs, chemistry, hematology, and urinalysis.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males or females between the ages of 18 to 55 years at Screening.
2. Body mass index between 18 kg/m2 to 33 kg/m2, inclusive, and body weight of >50 kg (110 pounds).
3. Female subjects must be surgically sterile (bilateral tubal ligation, hysterectomy, or bilateral oophorectomy at least 6 months prior to first study drug administration), at least two years post-menopausal, or willing to either (1) utilize hormonal contraception plus use one barrier method or (2) use two barrier methods of contraception from initial screening until one month after taking the final dose. Barrier methods of contraception include diaphragm, cervical cap, male condom, female condom, and spermicidal foam and sponges. An intrauterine device (IUD) is also considered a barrier method of contraception in this study; if the subject is using an IUD, she will need to use an additional barrier method of contraception. Menopausal status will be verified by testing for follicle stimulating hormone (FSH ≥25 mIU/mL) at Screening. In addition, all females must have a negative blood test for pregnancy within 28 days during the Screening period and negative urine test for pregnancy on Day-1 of each Treatment Visit regardless of childbearing potential.
4. Male subjects must be willing to inform female partners of their participation in the study and must agree to use adequate contraceptive methods (vasectomy performed at least 6 months prior to first study drug administration, or use at least one barrier method of birth control).
5. Able to understand the study procedures, voluntarily consent to participate in this study, and provide written informed consent prior to start of any study-specific procedures.
6. Willing and able to remain in the study unit for the required periods and return for each treatment of the six treatment periods, including the outpatient visits.

Exclusion Criteria:

1. Clinically significant abnormality, in the Investigator's judgement, in Screening hematology, chemistry, or urinalysis tests, or from medical history, social history, vital sign, or physical examination
2. Active liver disease or positive serology results for hepatitis B surface antigen (HbsAg), hepatitis C virus (HCV), or human immunodeficiency virus (HIV).
3. Abnormal liver function test at the Screening Visit (aspartate aminotransferase or alanine aminotransferase >2 × the upper limit of normal [ULN]; total bilirubin >1.5 × ULN; or alkaline phosphatase >2 × ULN based on appropriate age and gender normal values).
4. Current or past history of angle closure glaucoma, or diagnosis of angle closure glaucoma.
5. Marked hypotension (systolic blood pressure [BP] ˂90 mmHg or diastolic BP ˂50 mmHg) or hypertension (systolic BP ˃150 mmHg or diastolic BP ˃100 mmHg) based on sitting values obtained. Out-of-range results may be repeated once at Screening. This exclusion applies to the vital signs performed at Screening and on Day -1 on Treatment Period 1.
6. Marked bradycardia (heart rate ˂45 beats per minute [bpm]) or tachycardia (heart rate ˃110 bpm) based on supine ECG values obtained. Out-of-range results may be repeated once at Screening. This exclusion applies to the vital signs performed at Screening and on Day -1 on Treatment Period 1.
7. Current or past history of significant (in the Investigator's judgement) cardiovascular, cerebrovascular, pulmonary, renal, or liver disease. Stable, well-controlled hypertension and hyperlipidemias are allowed.
8. Clinically important or significant conduction abnormalities on single ECG or evidence or history of long QT syndrome based on supine ECG values obtained at Screening. Out-of-range results may be repeated once at Screening.
9. Current or past history of gastric or duodenal ulcers or other diseases of the gastrointestinal tract that could interfere with absorption of study drug. Note: Subjects with a history of appendectomy or cholecystectomy may be enrolled.
10. Active acute or chronic infectious diseases.
11. Unable to discontinue medications including anticholinergic agents, psychotropic drugs, sedative antihistamines, or other centrally active medications [e.g., CNS- penetrant beta blockers], and moderate to strong inhibitors or inducers of CYP3A4, CYP2D6, or other cytochromes) 14 days prior to the first dose of study drug (Period 1, Day 1) and during the study (Follow-Up). Other prescription or non-prescription drugs such as antihypertensive or cholesterol lowering drugs are allowed, if, in the Investigator's judgement, they would not interfere with the study medication or the cognitive testing.
12. Unable to discontinue and abstain from over-the-counter, herbal preparations, dietary supplements, nutraceuticals, vitamins and minerals at least 7 days prior to the first dose of study drug and during the study. The one exception to this rule is acetaminophen, which may be taken for minor ailments at doses up to 1000 mg per day.
13. Any history of alcohol or other substance abuse, including marijuana, within the previous year prior to the Screening visit (per the current edition of the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition: DSM-5), or regular (daily) consumption of alcohol exceeding two bottles of beer, or the equivalent amount of other forms of alcohol (1 serving = 12 oz beer, 5.0 oz wine, or 1.5 oz distilled spirits).
14. Any use of alcohol, grapefruit, marijuana, or other psychotropic agent within 12 hours of admission into the CRU.
15. Active smokers or tobacco users (e.g., chew and snuff) who are unable to discontinue tobacco use or nicotine-containing products (including e-cigarettes) at least 4 weeks prior to Screening and to refrain from using during the study.
16. Inability or unwillingness to comply with the protocol or likely inability to complete the study.
17. Participation in other clinical studies involving investigational drug within the previous 30 days prior to the Screening Visit.
18. Donation of blood within the prior 4 weeks, or blood products within the prior 2 weeks, prior to first study drug administration.
19. Positive result for drugs of abuse, alcohol, or cotinine at Screening, or a positive drug or alcohol (breath) result upon admission to CRU.
20. History of clinically significant drug allergy that includes symptoms such as shortness of breath, rash, or edema. This includes known hypersensitivity to donepezil hydrochloride, scopolamine, or belladonna, alkaloids.
21. Inability or unwillingness to perform the Cogstate cognitive function tests.
22. A suicidal ideation intensity score of 2 or higher per screening Columbia Suicide Severity Rating Scale (C-SSRS) assessment and/or any suicidal behavior within the past 28 days.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Groton Maze Learning Test (GMLT) | 2 hours post-scopolamine s.c. injection

OTHER OUTCOMES:
Detection Test (DET) | 30 minutes prior and at 1, 2, 3, 4, and 6 hours post-scopolamine sc injection
One Card Learning Test (OCL) | 30 minutes prior and at 1, 2, 3, 4, and 6 hours post-scopolamine sc injection
One Back Test (ONB) | 30 minutes prior and at 1, 2, 3, 4, and 6 hours post-scopolamine sc injection
Two Back Test (TWOB) | 30 minutes prior and at 1, 2, 3, 4, and 6 hours post-scopolamine sc injection
Physical exam, vital signs, clinical laboratory, ECG | Study duration up to 12 weeks
  To evaluate the safety and tolerability of BPN14770 in healthy subjects
Plasma concentrations of BPN14770 | Plasma BPN14770 concentrations at 0, 2.5, 4.5 and 6.5 hours post-scopolamine sc injection
  To obtain pharmacokinetic data on BPN14770

CONTACTS AND LOCATIONS:
Overall Officials: Cassandra Key, MD, Principal Investigator — ICON Early Phase Services, LLC
Locations (1):
- ICON Early Phase Services, LLC, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No